CLINICAL TRIAL: NCT02243397
Title: Molecular and Cellular Analysis of Breast Cancer
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Kathleen Horst, Kathleen Horst MD, Stanford University
Other Study IDs: IRB-29691
Record Dates: First submitted 2014-09-15; First posted 2014-09-17 (Estimated); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Breast - Female; Breast - Male

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, cerebrospinal fluid, abdominal fluid, chest fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the study is to investigate the different types and subtypes of cells found in breast tumors. The investigators will do this using a variety of molecular analysis tools that may allow for improved tests. The different types of cells in breast cancer impacts the way individuals respond to various treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven diagnosis of breast cancer or a carcinoma of unknown primary consistent with the presentation of a primary breast malignancy.
2. 18 years of age or older.
3. Ability to understand and the willingness to sign a written informed consent do

Exclusion Criteria:

* None

Min Age: 18 Minutes | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: breast cancer patients at Stanford Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 145 (Actual)
Dates: Start 2014-09-10 (Actual); Primary Completion 2021-04-19 (Actual); Study Completion 2021-04-19 (Actual)

PRIMARY OUTCOMES:
levels of GM-CSF in plasma | 10 years
  We will be measuring levels of GM-CSF (Granulocyte-macrophayge colony stimulating factor) from the plasma of the patient before during and after the irradiation treatment to study if there is any increase in the GM-CSF production

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Horst, Principal Investigator — Stanford University
Locations (1):
- Stanford University Cancer Institute, Stanford, California, United States